CLINICAL TRIAL: NCT07385794
Title: Design and Validation of a Personalized Preventive System for Adolescents Based on Biological Maturity, Body Composition, and Musculoskeletal Function.
Acronym: PREVEN-KID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Professor of Health Sciences, University of Alicante
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UA-2025-12-13; INNTA3/2025/8 (Other: Valencian Agency for Innovation)
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Health; Adolescent Growth and Development; Injury Prevention
Keywords: Adolescents; Biological maturation; Peak height velocity; Musculoskeletal function; Injury prevention; Physiotherapy; Preventive exercise; Physical development; Youth athletes

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either a personalized preventive physiotherapy and exercise intervention group or a usual activity control group, and followed in parallel with pre- and post-intervention assessments.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Preventive Physiotherapy Program (Experimental): Participants in this arm will receive a personalized preventive physiotherapy and exercise program tailored to their biological maturation status and functional profile. The intervention will last 12 weeks and will include two supervised sessions per week focusing on neuromuscular control, strength development, mobility, balance, and postural stability. Periodic reassessments will allow individualized progression and adjustment of the program throughout the intervention period.
  Interventions: Behavioral: Personalized Preventive Physiotherapy and Exercise Program
- Usual Activity Control Group (No Intervention): Participants in this arm will continue with their usual school and/or sports activities without receiving a structured preventive physiotherapy or exercise program. They will undergo the same baseline and post-intervention assessments as the intervention group for comparison purposes.

INTERVENTIONS:
Behavioral: Personalized Preventive Physiotherapy and Exercise Program — This intervention consists of a personalized preventive physiotherapy and exercise program designed according to each participant's biological maturation status and functional assessment. The program lasts 12 weeks and includes two supervised sessions per week. Sessions focus on neuromuscular control, strength development, mobility, balance, core stability, and postural control. The intervention is individualized based on baseline and periodic reassessments, allowing progression and adjustment throughout the program. All sessions are supervised by qualified professionals.
  Arms: Personalized Preventive Physiotherapy Program

SUMMARY:
This study aims to evaluate the effectiveness of a personalized preventive physiotherapy and exercise program based on biological maturation status in adolescents aged 14 to 15 years. During adolescence, rapid growth and differences in biological maturation can increase the risk of musculoskeletal imbalances, pain, and injuries, especially in physically active youth. However, most preventive programs are designed according to chronological age rather than biological development.

Participants will be assessed using non-invasive methods to determine biological maturation, body composition, and musculoskeletal function, including strength, balance, mobility, and postural control. Based on these assessments, participants in the intervention group will receive a 12-week individualized preventive physiotherapy program adapted to their maturation stage, while the control group will continue with their usual school or sports activities without structured intervention.

The study will compare changes in musculoskeletal function, body composition, pain perception, and lifestyle-related variables between baseline and post-intervention assessments. The results are expected to provide evidence for a maturation-based preventive approach that can be applied in clinical, school, and sports settings to reduce injury risk and improve musculoskeletal health in adolescents.

DETAILED DESCRIPTION:
Adolescence is a critical period of physical development characterized by rapid growth and significant interindividual variability in biological maturation. These changes can temporarily affect coordination, strength, and musculoskeletal balance, increasing the risk of pain, functional limitations, and sports-related injuries. Traditional preventive and training programs are commonly based on chronological age, which may not adequately reflect an adolescent's true biological development.

This study is a prospective, longitudinal, interventional study with a pre-post design and a non-randomized control group. A total of approximately 120 adolescents aged 14 to 15 years will be recruited from educational and sports institutions. Participants will be allocated to either an intervention group or a control group.

At baseline, all participants will undergo a comprehensive non-invasive assessment including anthropometry, estimation of biological maturation using validated predictive equations for peak height velocity, body composition analysis, and musculoskeletal function tests assessing strength, balance, mobility, and core stability. Subjective measures such as pain perception, sleep quality, physical activity level, and general well-being will also be collected using validated questionnaires.

Participants in the intervention group will complete a 12-week personalized preventive physiotherapy and exercise program, consisting of two supervised sessions per week. The program will be tailored to each participant's maturation status and functional profile, focusing on neuromuscular control, mobility, strength development, and postural stability. Periodic reassessments will allow for individualized progression and adjustment of the intervention. The control group will continue with their usual routines without receiving a structured preventive program.

Post-intervention assessments will replicate baseline measurements to evaluate changes over time. The primary outcomes will include changes in musculoskeletal function parameters, while secondary outcomes will assess body composition, pain perception, lifestyle variables, and adherence to the intervention.

The findings of this study aim to support the use of biologically informed preventive strategies in adolescents and to contribute to the development of scalable, evidence-based programs for clinical, educational, and sports environments.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 14 to 15 years at the time of enrollment.
* Male and female participants.
* Apparently healthy adolescents without diagnosed chronic medical conditions.
* Participation in regular school physical education and/or organized sports activities.
* Ability to participate in moderate physical activity as determined by a pre-participation screening.
* Written informed consent obtained from parents or legal guardians, and assent from the participant.

Exclusion Criteria:

* Presence of acute or chronic musculoskeletal injury that limits participation in physical activity at the time of enrollment.
* History of musculoskeletal surgery within the previous 12 months.
* Diagnosed neurological, cardiovascular, metabolic, or systemic disease that contraindicates physical exercise.
* Current participation in another structured exercise or intervention study.
* Use of medication that may significantly affect musculoskeletal function or physical performance.
* Any condition that, in the opinion of the investigators, could compromise participant safety or adherence to the protocol.

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Lower-limb Strength (Isometric) | Baseline and 12 weeks
  Change in lower-limb isometric strength assessed using digital dynamometry during standardized testing procedures.
Postural Balance | Baseline and 12 weeks
  Change in postural balance assessed using instrumented balance testing (e.g., force platform and inertial sensors) during standardized static and dynamic tasks.

SECONDARY OUTCOMES:
Mobility / Range of Motion | Baseline and 12 weeks
  Change in joint mobility assessed as active range of motion using motion sensors or standardized mobility tests.
Postural Control | Baseline and 12 weeks
  Change in postural control parameters derived from instrumented postural assessment (e.g., center of pressure metrics and/or inertial sensor outputs) during standardized tasks.
Core Stability / Core Control | Baseline and 12 weeks
  Change in core stability assessed using a standardized core control test protocol (e.g., ICAROS-based assessment).
Vertical Jump Performance | Baseline and 12 weeks
  Change in vertical jump performance assessed using squat jump and/or countermovement jump measured with a load cell or force platform.
Fat Mass | Baseline and 12 weeks
  Change in fat mass assessed using multi-frequency bioelectrical impedance analysis and/or anthropometric assessment, following standardized procedures.
Skeletal Muscle Mass | Baseline and 12 weeks
  Change in skeletal muscle mass and/or fat-free mass assessed using multi-frequency bioelectrical impedance analysis, following standardized procedures.
Phase Angle | Baseline and 12 weeks
  Change in phase angle derived from multi-frequency bioelectrical impedance analysis.
Maturity Offset | Baseline and 12 weeks
  Change in maturity offset estimated using validated anthropometric equations.
Peak Height Velocity (PHV) Status | Baseline and 12 weeks
  Change in estimated PHV status (pre-, circa-, post-PHV) derived from validated predictive equations.
Musculoskeletal Pain Intensity | Baseline and 12 weeks
  Change in self-reported musculoskeletal pain intensity assessed using a standardized pain rating scale.
Physical Activity Level (PAQ-A) | Baseline and 12 weeks
  Change in physical activity level assessed using the Physical Activity Questionnaire for Adolescents (PAQ-A).
Sleep Quality | Baseline and 12 weeks
  Change in self-reported sleep quality assessed using a standardized questionnaire.
Intervention Adherence | Baseline and 12 weeks
  Adherence measured as the percentage of completed supervised sessions out of the total prescribed sessions during the 12-week intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- European Institute of Exercise and Health, Alicante, Elche, Spain

IPD SHARING:
Plan to Share IPD: No